CLINICAL TRIAL: NCT01675336
Title: The Association Between Interleukin-1 Gene Variations and Adult Chronic Periodontal Disease in Chinese (Taiwan))
Brief Title: Genetics of Periodontal Diseases in Chinese (Taiwan)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University (Other)
Collaborators: Interleukin Genetics, Inc. (Industry)
Responsible Party: Principal Investigator, Ya-Ping Ho, Assistant Professor, Kaohsiung Medical University
Other Study IDs: ILI-11-129-PST2Taiwan
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective case control study to validate the association between Interleukin-1 gene variations and adult chronic periodontal disease in Chinese (Taiwan).

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, an individual needs to be Han Chinese of 35 years of age or older at time of enrollment.

Exclusion Criteria:

* Subjects who, at time of enrollment, were pregnant or breastfeeding, or needed antibiotic prophylaxis before periodontal treatment will be excluded from this study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All study subjects will be selected from a pre-existing patient database in Taiwan. All chronic periodontitis cases and controls will be subjects who were at least 35 years old at time of enrollment.
  Classification of chronic periodontitis will be based on the extent of periodontal tissue destruction with consideration of tooth loss.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-08

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ping Ho, Ph.D., Principal Investigator — employee